CLINICAL TRIAL: NCT03307213
Title: Evaluation of the Efficacy (QCA) and Safety of the BioFreedom™ Biolimus A9™ CoCr Stent in a Randomised Trial in Patients With CAD
Brief Title: BioFreedom QCA Study in CAD Patients
Acronym: BioFreedomQCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17EU02
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease; Cardiac Death; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Death; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to one of the treatment arms to receive either the BioFreedom™ SS or the BioFreedom™ CoCr stent.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioFreedom™CoCr (Experimental): Patients with CAD will receive the BioFreedom™CoCr stent if randomised to this arm.
  Interventions: Device: BioFreedom™ CoCr Biolimus A9™ stent
- BioFreedom™ SS (Active Comparator): Patients with CAD will receive the BioFreedom™SS stent if randomised to this arm.
  Interventions: Device: BioFreedom™ SS Biolimus A9™ stent

INTERVENTIONS:
Device: BioFreedom™ CoCr Biolimus A9™ stent — Stent implantation
  Arms: BioFreedom™CoCr
Device: BioFreedom™ SS Biolimus A9™ stent — Stent implantation
  Arms: BioFreedom™ SS

SUMMARY:
This study aims to demonstrate that the BioFreedom™ Cobalt Chromium Drug Coated Stent is non-inferior to the market authorized BioFreedom™ Stainless Steel Stent with respective to efficacy and shows a similar safety profile.

DETAILED DESCRIPTION:
The BioFreedom™ QCA trial is designed to evaluate the safety and efficacy of the BioFreedom™ CoCr DCS coronary stent system compared to the Biofreedom™ stainless steel DCS coronary stent system, in a randomized controlled trial on an all-comers patient population.

The primary objective is to measure non-inferiority of the BioFreedom™ CoCr stent compared to BioFreedom™ DCS as measured by the difference in angiographically measured late lumen loss at 9 months, and the main secondary endpoint is to assess safety as measured by MACE and ST. Two hundred (200) patients will be randomized 1:1 to either stent, allowing for a direct comparison, and will be followed-up to 2 years to measure for late MACE and ST events.

ELIGIBILITY:
Inclusion Criteria:

"Real world, all comer" patients

1. Age ≥18 years;
2. Symptomatic coronary artery disease including patients with chronic stable angina, unstable angina, silent ischemia, and acute coronary syndromes including non-ST elevation myocardial infarction and ST-elevation myocardial infarction;
3. Presence of one or more coronary artery stenosis >50% in a native coronary artery or a saphenous bypass graft from 2.50 to 3.5 mm in diameter that can be covered with one or multiple stents (angiographic inclusion);
4. No limitation on the number of treated lesions, and vessels, and lesion length

Exclusion Criteria:

1. Individual is pregnant, nursing or planning to be pregnant;
2. Known intolerance to aspirin, clopidogrel, heparin, stainless steel, cobalt chromium, Biolimus A9™ or contrast material
3. Inability to provide informed consent;

Note: Not all exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
In-stent late lumen loss (LLL) at 9 months | 9 months
  In-stent late lumen loss (LLL) assessed by quantitative coronary angiography (QCA) at 9 months

SECONDARY OUTCOMES:
Cardiac Death | 1, 9, 12 and 24 months
  Cardiac Death
Myocardial infarction | 1, 9, 12 and 24 months
  Myocardial infarction
MACE | 1, 9, 12 and 24 months
  MACE defined as cardiac death, myocardial infarction and clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Manel Sabate, Dr., Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No